CLINICAL TRIAL: NCT07016347
Title: Elevated Plasma GDF15 Combined With FGF21 Suggests Mitochondrial Dysfunction in a Subgroup of Anorexia Nervosa Patients
Brief Title: GDF15 in Anorexia Nervosa
Status: Completed | Type: Observational
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Ida AK Nilsson, Principal investigator, Karolinska Institutet
Other Study IDs: GDF15 in AN
Record Dates: First submitted 2025-05-21; First posted 2025-06-11 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-03

CONDITIONS: Anorexia Nervosa
MeSH Terms: conditions — Anorexia Nervosa

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- active anorexia nervosa
- recovered anorexia nervosa
- healthy controls

SUMMARY:
Evaluating plasma levels of a protein called GDF15 in active and recovered anorexia nervosa, as well as healthy controls

ELIGIBILITY:
Inclusion Criteria:

- active DSMV diagnosis of anorexia nervosa/ at least two years of recovery from DSMV anorexia nervosa / no history of anorexia nervosa

Exclusion Criteria:

- male

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: swedish population
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2017-01-23 (Actual); Primary Completion 2021-11-15 (Actual); Study Completion 2024-11-04 (Actual)

PRIMARY OUTCOMES:
plasma GDF15 | At baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Karolinska Institutet, Stockholm, Sweden